CLINICAL TRIAL: NCT04066296
Title: A Double Blinded Randomized Control Trial in Outcomes for Lumbar Decompressions With Use of Liposomal Bupivicaine
Brief Title: Outcomes for Lumbar Decompressions With Use of Liposomal Bupivicaine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-0903
Record Dates: First submitted 2019-07-03; First posted 2019-08-26 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The PI, co-Investigators, and clinicians will be blinded to the patient's treatment arm. The pharmacist will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivicaine (Active Comparator): Treatment with liposomal bupivicaine
  Interventions: Drug: Liposomal bupivacaine
- Standard Local Anesthestic (Active Comparator): Treatment with Standard Local Anesthestic
  Interventions: Drug: Liposomal bupivacaine

INTERVENTIONS:
Drug: Liposomal bupivacaine — Injection of either liposomal bupivicaine or standard local anesthetic during surgical procedure.
  Other Names: standard local anesthetic

SUMMARY:
Evaluate the benefit of using liposomal bupivicaine in lumbar laminectomies in terms of length of stay, IV narcotic use, 30-day narcotic use, visual analog score (VAS) and 30-day readmissions

DETAILED DESCRIPTION:
Recent evidence suggests the use of liposomal bupivicaine (LB) in lumbar spine surgery shortens length of hospital stay and overall post-operative narcotic use. Studies have shown its utility in single level microdiscectomies and lumbar fusions, but there have been no publications regarding lumbar laminectomies and associated outcomes with LB. The investigators' hypothesis is that LB will significantly shorten inpatient stays as well as overall narcotic usage in single, double or multi-level lumbar laminectomies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Adult (≥18 yo)
3. Lumbar stenosis

Exclusion Criteria:

1. Co-morbidities precluding surgery
2. ≤18 yo
3. Pregnant
4. Breastfeeding
5. Need for instrumented fusion
6. Prisoners
7. Intra-operative CSF leak (identified by gush of CSF)
8. Daily pre-operative opioid use of > 25 morphine Eq/day
9. Previous lumbar surgery at indicated level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Overall length of hospital stay from hospital admission to hospital discharge | From date of hospital admission until date of hospital discharge, assessed up to 2 weeks.
  Length of stay will be measured in hours

SECONDARY OUTCOMES:
IV narcotic usage | From date of hospital admission until date of hospital discharge, assessed up to 2 weeks.
  Tracked by patient's electronic medical record
30-day narcotic usage | 30-day post surgery
  Narcotic usage will be assessed via state narcotic databases.
Change in Visual Analog Pain scale scores | Screening, Day of Procedure, Prior to Hospital Discharge (Post-op, Up to 2 weeks), Up to 30-days post-surgery (Follow-Up#1) and up to 12-months post-op follow up
  The scale is called the Visual Analog Pain scale. This scale provides a measure of the patient's reported level of pain . Patients will be asked to rate their pain level using the Visual Analog Pain scale. This scale uses numbers, 1-10, with 1 being no pain and 10 being the worst pain. It also uses faces depicting no pain up to the worst pain. Lower reported scores indicate the patient has little to no pain, which is desirable.
30-day readmission rates | Day 30
  Occurrences of readmission will be tracked by patient's electronic medical record

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.